CLINICAL TRIAL: NCT07008885
Title: A Phase I/II Single-center Study Evaluating the Safety and Efficacy of BCOR and ZC3H12 Genes Knock-out CD19-targeting CAR-T Cell Therapy in Adults With Refractory/Relapsed B-cell Acute Lymphoblastic Leukaemia
Brief Title: BCOR and ZC3H12 Genes Knock-out CD19-targeting CAR-T Cell Therapy in r/r B-ALL
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Han weidong, Director of Biotherapeutic Department, Chinese PLA General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CHN-PLAGH-BT-090
Record Dates: First submitted 2025-05-21; First posted 2025-06-06 (Actual); Last update posted 2025-06-25 (Actual); Status verified 2025-06

CONDITIONS: Acute Lymphocytic Leukemia
Keywords: CAR-T cells; ALL; CD19
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — fludarabine; fludarabine phosphate; Injections; Cyclophosphamide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CAR19TIF cells (Experimental): Patients with r/r B-ALL A conditioning chemotherapy regimen of fludarabine and cyclophosphamide will be administered followed by investigational treatment, CAR19TIF cells.
  Interventions: Biological: CAR19TIF cells; Drug: Fludarabine; Drug: Cyclophosphamide

INTERVENTIONS:
Biological: CAR19TIF cells — Phase 1 dose escalation/decline (3+3) :
  starting dose: 5×10^5 cells/kg, According to effective expansion and clinical efficacy data, a descending dose escalation model will be adopted: such as 1×10^5 cells/kg, 5×10^4 cells/kg.
  If the 5×10^5 cells/kg dose group does not achieve efficient expansion and clinical benefit, an ascending dose escalation model will be adopted, such as 2×10^6 cells/kg, 6×10^6 cells/kg.
  Phase 2 : dose of RP2D.
  Other Names: BCOR and ZC3H12 genes knock-out CD19 CAR T cells
Drug: Fludarabine — Intravenous fludarabine 25~30 mg/m^2/day on days
  -5, -4, and -3.
  Other Names: Fludarabine Phosphate for Injection
Drug: Cyclophosphamide — Intravenous cyclophosphamide 250~500 mg/m^2/day on days -5, -4, and -3.
  Other Names: Cyclophosphamide for Injection

SUMMARY:
In this single-center, single-arm, prospective, Phase 1/2 study, the safety and efficacy of autologous BCOR and ZC3H12 genes knock-out CD19-targeting chimeric antigen receptor (CAR) T-cell therapy will be evaluated in patients with refractory/relapsed (r/r) B-cell acute lymphoblastic leukaemia (B-ALL).

In phase 1, 3 eligible patients will be enrolled and receive BCOR and ZC3H12 genes knock-out CD19 CAR T cell therapy at a initial dose of 5×10^5 cells/kg. Based on the results, . Subsequently an additional 3-15 patients will be enrolled in a "3+3" dose-escalation/decline design to adjust the dose of BCOR and ZC3H12 genes knock-out CD19 CAR T cells to achieve optimal safety and efficacy. The recommended Phase 2 dose (RP2D) will then be established. 10 to 12 subjects will be enrolled and receive BCOR and ZC3H12 genes knock-out CD19 CAR T cell infusion at dose of RP2D.

DETAILED DESCRIPTION:
CAR T-cell therapy targeting CD19 has transformed the management of r/r B-ALL, complete remission (CR) or complete response with incomplete count recovery (CRi) has been achieved as many as 70-90% in r/r B-ALL cases. Unfortunately, 40-60% of patients responding to this therapy relapse within 1 year due to challenges such as limited CAR T cell persistence,T cell exhaustion,etc. These limitations highlighted the need for further optimization of the CAR T cell design to improve the efficiency of CD19-targeted CAR T cell therapy in r/r B-ALL.

The investigators have developed that the suppression of two genes, Zc3h12a and Bcor, induced CD19 CAR T cells capable of expansion, persistence, and inducing long-term B cell depletion in immunocompetent mice models,even without any conditioning and in low dose infusion. From this, the investigators present a single-center, single-arm, prospective, phase 1/2 study to evaluate the safety and efficacy of BCOR and ZC3H12 genes knock-out CD19 CAR T cells in adult patients with r/r B-ALL. For simplicity, the investigators have termed these CD19 CAR T cells lacking ZC3H12A and BCOR as immortal-like and functional CD19 CAR T (CAR19TIF) cells, reflecting their immortal-like and functional characteristics.

Phase 1 (dose escalation/decline)

In phase 1, 6-18 subjects will be enrolled. Referring to the starting dose of most CAR T cell therapies, and to avoid exposing patients to the risk of "ineffective expansion dose", 3 patients will receive CAR19TIF cells therapy at a starting dose of 5×10^5 cells/kg.According to the copy number of CAR T cells were assessed by number in peripheral blood and clinical efficacy data, additional 3-15 patients will be enrolled in a "3+3" dose-escalation/decline design to adjust the dose of CAR19TIF cells to achieve optimal safety and efficacy :

After obtaining effective expansion data and clinical efficacy data, a descending dose escalation model will be adopted: such as 1×10^5 cells/kg, 5×10^4 cells/kg. If the 5×10^5 cells/kg dose group does not achieve efficient expansion and clinical benefit, an ascending dose escalation model will be adopted, such as 2×10^6 cells/kg, 6×10^6 cells/kg.

3 subjects are enrolled in a cohort corresponding to a dose level. If 1 subject in a cohort of 3 subjects experiences a DLT, 3 additional subjects will be enrolled at the current dose level.

For safety purposes, the administration of CAR19TIF cells will be staggered by 28 days between the first two subjects in each cohort. And for each of the remaining cohorts, the administration of CAR19TIF cells will be staggered by 28 day.

Phase 2 (expansion cohort) In phase 2, 10 to 12 subjects will be enrolled and receive cell infusion at dose of RP2D, which will be determined based on the maximum tolerated dose (MTD), occurrence of DLT, the obtained efficacy results, pharmacokinetics/pharmacodynamics and other data according to the phase 1.

Objectives The primary objectives of the phase 1 were to evaluate the tolerability and safety of CAR19TIF cells in patients with r/r B-ALL, and determine RP2D. The primary purpose of the phase 2 study was to evaluate the efficacy of CAR19TIF cells n the above population.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-70 (inclusive),gender unrestricted.
2. Patient with r/r CD19+ B-ALL, as per guidelines (NCCN, 2019)

   * morphologically confirmed with ≥ 5% leukaemic blasts in the bonemarrow;
   * or presenting a quantifiable MRD load of 1x10^-3 , assessed by multiparameter flow cytometry and/or quantitative polymerase chain reaction, at the end of the last induction treatment.
   * who has exhausted alternative treatment options.

   Relapsed disease is defined as:
   * second or subsequent bone marrow relapse or,
   * any bone marrow relapse after allogenic hematopoiesis stem cell transplant (allo-HSCT).

   Refractory disease is defined by not achieving an initial complete response (CR) after 2 cycles of a standard chemotherapy regimen (primary refractory). Subjects who were refractory to subsequent chemotherapy regimens after an initial remission were considered chemorefractory.
3. Toxicities due to prior therapy must be stable and recovered to ≤ Grade 1 (except for hematological toxicities and clinically non-significant toxicities such as alopecia).
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Adequate renal, hepatic, pulmonary and cardiac function defined as:

   * Serum creatinine≤1.5 upper limit of normal (ULN) or creatinine clearance (as estimated by Cockcroft Gault) ≥ 60 mL/min.
   * Serum alanine aminotransferase / aspartate aminotransferase (ALT/AST) ≤ 3×ULN; Total bilirubin ≤ 1.5×ULN.
   * Cardiac ejection fraction ≥ 50%, no evidence of pericardial effusion as determined by an echocardiogram (ECHO), and no clinically significant electrocardiogram (ECG) findings.
   * Coagulation Function: International Normalized Ratio (INR) ≤ 1.5 ×ULN, and Activated Partial Thromboplastin Time (APTT) ≤ 1.5×ULN .• Baseline oxygen saturation >91% on room air.
6. Subjects of both genders who are willing to practice birth control from the time of consent through 6 months after the completion of conditioning chemotherapy. Females of childbearing potential must have a negative serum or urine pregnancy test (females who have undergone surgical sterilization or who have been postmenopausal for at least 2 years are not considered to be of childbearing potential).
7. Voluntarily participate in this clinical trial and sign an informed consent form.

Exclusion Criteria:

1. Expected survival time < 3 months per Principal Investigator's opinion.
2. Previous or concurrent cancer within 3 years prior to treatment start EXCEPT for curatively treated cervical cancer in situ, non-melanoma skin cancer, superficial bladder tumors [Ta (non-invasive tumor), Tis (carcinoma in situ) and T1 (tumor invades lamina propria)].
3. Prior CD19 targeted therapy
4. Prior CAR-T therapy or other genetically modified T cell therapy.
5. Active central nervous system (CNS) leukaemia (CNS-3).
6. B-ALL with clinically suspected extra-medullary involvement.
7. Burkitt cell (L3 ALL) or mixed lineage acute leukaemia.
8. Clinically active significant CNS dysfunction

   * History or presence of CNS disorder such as seizure disorder, cerebrovascular ischemia/hemorrhage, dementia, cerebellar disease, or any autoimmune disease with CNS involvement.
   * Known history of irreversible severe neurological toxicity related to previous antileukaemic treatment leading to organic central nervous system lesions.
   * Radioimmunotherapy, radiotherapy, within 8 weeks (except prophylaxis of CNS involvement) before Inclusion.
9. Use of previous anti-leukemic therapy within 5 half-lives prior to CAR19TIF cells administration; participation in non-interventional registries or epidemiological studies is allowed.
10. History of severe, immediate hypersensitivity reaction attributed to lymphodepletion drugs or any component of CAR19TIF cells.
11. Presence or suspicion of fungal, bacterial, viral, or other infection that is uncontrolled or requiring intravenous (IV) antimicrobials for management.
12. Uncontrolled or active infectious diseases, such as human immunodeficiency virus (HIV) infection, acute or chronic active hepatitis B or C, epstein-barr virus (EBV), and cytomegalovirus (CMV) infection.
13. Subjects with cardiac atrial or cardiac ventricular lymphoma involvement.
14. History of myocardial infarction, cardiac angioplasty or stenting, unstable angina, or other clinically significant cardiac disease within 12 months of enrollment.
15. Expected or possible requirement for urgent therapy within 6 weeks due to ongoing or impending oncologic emergency (eg, tumor mass effect, tumor lysis syndrome).
16. Primary immunodeficiency.
17. History of autoimmune disease (e.g. Crohn's, rheumatoid arthritis, systemic lupus) resulting in end organ injury or requiring systemic immunosuppression/systemic disease modifying agents within the last 2 years.
18. History of symptomatic deep vein thrombosis or pulmonary embolism requiring systemic anticoagulation within 6 months of enrollment.
19. Any medical condition likely to interfere with assessment of safety or efficacy of study treatment.
20. Vaccine ≤ 6 weeks prior to planned start of conditioning regimen.
21. In the investigator's judgment, the subject is unlikely to complete all protocol-required study visits or procedures, including follow-up visits, or comply with the study requirements for participation.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2027-05-31 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Incidence of Adverse Events (AEs) | Up to 12 months since the initiation of CAR-T cell therapy.
  AE is defined as any adverse medical event from the date of randomization to 12 months after CAR T cells infusion. Among them, cytokine release syndrome(CRS) and immune cell-associated neurotoxicity syndrome (ICANS) were graded according to American Society for Transplantation and Cellular Therapy (ASTCT) criteria. Other AEs were graded according to common terminology criteria for adverse events (CTCAE) v5.0.
Phase 1:Incidence of Incidence of Dose-Limiting Toxicities (DLTs) | [Time Frame: Up to 28 days since the initiation of CAR-T cell therapy]
  DLT is defined as any AE related to the investigational drug that occurs within 28 days after administration of the CAR19TIF cells and meets any one of the criteria listed in the DLT criteria:
  * Grade 3 CRS that does not resolve to grade 2 or lower within 2 weeks;
  * Grade 3 ICANS lasting for ≥ 7 days;
  * Any Grade ≥ 4 CRS or ICANS;
  * Any other Grade ≥ 4 and Grade 3 AEs related to the CAR19TIF cells that lasts for ≥ 14 days, except hematology toxicity.
Phase 1:RP2D | 12 months
  The recommended dose for phase 2 was determined through phase 1 study.
Phase 2:Objective response rate (ORR) | 24 months
  Objective response definition: a molecular response (MRD < 10^-4 post treatment) assessed by multiparameter flow cytometry and/or qPCR, or a morphologic complete response (CR), or a CR with incomplete blood count recovery (CRi). ORR is defined as the proportion of patients who have achieved objective response assessed by investigators.
Phase 2:Overall Survival (OS) | 24 months
  OS is defined as the time from CAR-T cells infusion to the date of death. Subjects who have not died by the analysis data cutoff date will be censored at the last contact date.
Phase 2: Progression Free Survival (PFS) | 24 months
  PFS is defined as the time from the CAR-T cells infusion date to the date of disease progression assessed by investigators, or death any cause. Participants not meeting the criteria for progression by the analysis data cutoff date were censored at the last evaluable disease assessment date.

SECONDARY OUTCOMES:
Phase 1 and phase 2: Level of CAR-positive T cells circulating in blood over time | 12 months
  Number and copy number of CAR-T cells were assessed by number in peripheral blood. Blood samples were collected before and one year after cell infusion (until CAR-T cells were not detected for two consecutive times) to detect the number and copy number of CAR-T cells, and to evaluate the pharmacokinetics of CAR-T.
Phase 1 and phase 2: Level of CD19+ cells in peripheral blood | 12 months
  The level of CD19+ cells in peripheral blood will be detected by flow cytometry.

OTHER OUTCOMES:
Relationship between infusion dose of CAR T cells and efficacy. | 24 months
  Peripheral blood was collected at the day of infusion (day 1), day 4, day 7, day 11, day 14, day 28, at least once every month after 28 days, at least once every three months after half a year, and at least once every six months after a year. The researchers will analyze the relationship between the number of CAR T cells, copy number, cytokines level, and efficacy of CAR T cells. The number of CAR T cells was detected by flow cytometry, and the copy number was detected by quantitative PCR (qPCR).
To analyze the dynamic changes of CAR T cells after infusion | 24 months
  he dynamic changes of the number (cells/ul)and copy number (copies/ug DNA) of CAR T cells in patients after CAR T treatment were analyzed. To summarize the characteristic of the peak(cells/ul) , expansion pattern, continuous expansion time (days )and evolution of CAR T cells in vivo.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Han, Ph.D, Principal Investigator — Biotherapeutic Department, Chinese PLA General Hospital
Locations (2):
- China (2):
  - China, Beijing, Biotherapeutic Department of Chinese PLA General Hospital
  - China, Beijing, Biotherapeutic Department of Chinsese PLA Gereral Hospital